CLINICAL TRIAL: NCT03263416
Title: Regional, Multicentric, Randomized Study Evaluating Treatment Adherence in Patients Treated With Oral Targeted Therapy in Oncology Supported by a Dedicated and Coordinated Follow-up (Using a Telephone Follow-up by a Nurse and a Pharmaceutical Conciliation) Compared to Standard Follow-up.
Brief Title: Study Evaluating Treatment Adherence in Patients Treated With Oral Targeted Therapy in Oncology Supported by a Dedicated and Coordinated Follow-up Compared to Standard Follow-up.
Acronym: ADHESIPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17GENE02
Record Dates: First submitted 2017-08-04; First posted 2017-08-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Solid Tumor
Keywords: Metastatic solid tumor; Oral Targeted Therapy; Treatment adherence
MeSH Terms: conditions — Neoplasm Metastasis; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Other: Dedicated and coordinated follow-up
- Arm B (Other): Standard
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: Dedicated and coordinated follow-up — * Coordinated follow-up performed by a dedicated nurse with consultations (before treatment initiation and during treatment) and a telephone follow-up during treatment period
  * Pharmaceutical conciliation before treatment initiation made by the Center Pharmacist
  * Completion of QLQ-C30 and GIRERD questionnaires
  Arms: Arm A
Other: Standard follow-up — - Completion of QLQ-C30 and GIRERD questionnaires
  Arms: Arm B

SUMMARY:
This is a prospective, comparative, open label, randomized, multicentric study evaluating the benefit of a dedicated and coordinated follow-up on treatment adherence in patients with metastatic solid tumor and starting a first cycle of treatment compared to standard follow-up. A dedicated and coordinated follow-up during the treatment period will be based on a telephone follow-up and a pharmaceutical conciliation.

Patients will be randomized into one of two study arms:

Arm A (Experimental follow-up): coordinated follow-up performed by a dedicated nurse and a pharmaceutical conciliation made by the Center Pharmacist.

Arm B: Standard follow-up during the treatment period.

Patients will be followed during 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a metastatic solid tumor and starting a first cycle of oral targeted therapy whatever the treatment line
2. Age > or = 18 years old
3. Affiliated to the french social security system
4. Patient must provide written informed consent prior to any study-specific procedure or assessment

Exclusion Criteria:

1. Patient not available by phone or with no caregiver who can answer the phone for him
2. Pregnant or breastfeeding women
3. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
4. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Efficacy: rate of patients who adhere to oral targeted therapy treatment administration. | 6 months per patient
  This outcome will be assessed by the counting of tablets and the completion of the GIRERD questionnaire by the patient (assessment performed at 1, 3 and 6 months during the treatment)

SECONDARY OUTCOMES:
Evaluation of the number of drug adaptations proposed by the Center Pharmacist following the pharmaceutical conciliation | 6 months per patient
Quality of life using the QLQ-C30 questionnaire | 6 months per patient
Safety according to the classification of the Common for Toxicity Criteria for Adverse Events (CTCAE) V4.03 | 6 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHEVREAU, MD, Principal Investigator — Institut Universitaire du Cancer Toulouse Oncopole
Locations (4):
- France (4):
  - Clinique Claude Bernard, Albi
  - Centre Hospitalier Intercommunal Castres Mazamet, Castres
  - Clinique Des Cedres, Cornebarrieu
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No